CLINICAL TRIAL: NCT05376722
Title: A Prospective Clinical Study of the Safety and Efficacy of Pamiparib Combined With Abiraterone Acetate in Neoadjuvant Treatment of High-risk or Very High-risk Localized Prostate Cancer
Brief Title: A Study of Pamiparib Combined With Abiraterone Acetate in Neoadjuvant Treatment of Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hongqian Guo (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); The First Affiliated Hospital of Soochow University (Other); Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor-Investigator, Hongqian Guo, Chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-PC-111
Record Dates: First submitted 2022-02-23; First posted 2022-05-17 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-10

CONDITIONS: Neoadjuvant Therapy
Keywords: pamiparib; abiraterone acetate; high-risk prostate cancer
MeSH Terms: interventions — pamiparib; abiraterone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pamiparib (Experimental): Subjects received pamiparib 40 mg orally, twice a day; abiraterone acetate 1000 mg orally, once a day; prednisone acetate tablets (prednisone) 5 mg, once a day; every 30 days Treatment cycle, treatment for 4-6 cycles, that is, 4-6 months. Robot-assisted laparoscopic radical prostatectomy and extended lymph node dissection within 30 days of the end of 4 months of neoadjuvant therapy. If the subjects have intolerable toxic reactions during the treatment period, the dose adjustment can be carried out. Day 1 of cycle 1, day 15 and day 1±3 days of each cycle thereafter, and 1 follow-up within 30 days after the end of treatment and before surgery; 1 prostate MRI during the screening period and within 30 days after the end of treatment and before surgery Scan, PSMA PET/CT scan or CT scan
  Interventions: Drug: pamiparib; Drug: abiraterone; Drug: prednisone

INTERVENTIONS:
Drug: pamiparib — pamiparib 40 mg orally, twice a day
Drug: abiraterone — biraterone acetate 1000 mg orally, once a day
Drug: prednisone — prednisone acetate tablets (prednisone) 5 mg, once a day

SUMMARY:
To evaluate the pathological response rate of pamiparib combined with abiraterone acetate in neoadjuvant therapy for surgically resectable high-risk or very high-risk prostate cancer after radical prostatectomy

DETAILED DESCRIPTION:
the main purpose: To evaluate the pathological response rate of pamiparib combined with abiraterone acetate in neoadjuvant treatment of surgically resectable high-risk or very high-risk prostate cancer after radical prostatectomy; Note: pathological response rate = pathological complete response rate (pCR) + minimal residual disease (MRD)(defined as residual tumor with the largest crosssection dimension ≤5 mm OR RCB≤0.25CM³)

Secondary purpose:

1. To evaluate the safety of pamiparib combined with abiraterone acetate as neoadjuvant therapy for high-risk or very high-risk prostate cancer;
2. To evaluate the rate of PSA biochemical recurrence-free survival (bPFS) at 1 year after radical prostatectomy in neoadjuvant treatment of high-risk or very-high-risk prostate cancer with pamiparib combined with abiraterone acetate;
3. The positive rate of surgical margins in radical prostatectomy;
4. Downstaging rate of radical prostatectomy;
5. Pathological response rate of neoadjuvant patients with HRR gene mutation;

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Men aged ≥18 years and ≤80 years old.
  2. Patients with prostate cancer diagnosed by histology or cytology who are suitable for radical prostatectomy.
  3. All patients meet at least one of the following criteria:

     1. Multiparametric MRI and PSMA PET/CT scan or CT scan showing primary tumor stage ≥ T3;
     2. Primary tumor Gleason score ≥ 8;
     3. Serum PSA concentration ≥ 20 ng/ml;
     4. Imaging assessment has regional lymph node metastasis (N1);
  4. Eastern Cooperative Oncology Group (ECOG) performance status score≤1
  5. Laboratory inspections meet the following requirements:

     Blood routine: white blood cell count (WBC) ≥3.0×109/L, platelet count ≥100×109/L, hemoglobin ≥9g/dl; renal function: serum creatinine ≤2×ULN; liver function: alanine aminotransferase (ALT) and Aspartate aminotransferase (AST)≤2.5×ULN, total bilirubin TBIL≤1.5×ULN; coagulation function: international normalized ratio (INR)<1.5.
  6. The subjects participate voluntarily, and the subjects themselves must sign the Informed Consent Form (ICF), indicating that they understand the purpose and required procedures of this research, and are willing to participate in the research. Subjects must be willing and comply with the prohibitions and restrictions set forth in the study protocol.
  7. During the treatment, the testosterone level in the blood is reduced to the "castration" level, and the testosterone level is less than 50ng/dL;
  8. The subjects can understand and are willing to sign the informed consent

Exclusion Criteria:

* Exclusion Criteria:

  1. Patients with neuroendocrine, small cell, or sarcomatoid features on prostate histopathology.
  2. Low- and intermediate-risk localized prostate cancer (all the following conditions are met) (PSA<20 ng/mL; Gleason score<8; clinical stage<T3).
  3. Patients with clinical or radiological evidence suggestive of extraregional lymph node metastasis or bone or visceral metastasis (any M1).
  4. Received androgen deprivation therapy (including drug or surgical castration) for more than 3 months or focal prostate cancer treatment or prostate cancer radiotherapy and chemotherapy in the past.
  5. Patients with severe or uncontrolled concurrent infections.
  6. Suffering from New York Heart Association (NYHA) class III/IV congestive heart failure, unstable angina or a history of myocardial infarction within the past 6 months.
  7. Uncontrolled severe hypertension, persistent uncontrolled diabetes, oxygen-dependent lung disease, chronic liver disease, or HIV infection.
  8. In the past 5 years, other malignancies other than prostate cancer, but cured basal or squamous cell skin cancer can be enrolled.
  9. Suffering from mental illness, mental disability or inability to give informed consent.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
the pathological response rate of pamiparib combined with abiraterone acetate in neoadjuvant therapy for surgically resectable high-risk or very high-risk prostate cancer after radical prostatectomy | up to 6months
  To evaluate the pathological response rate of pamiparib combined with abiraterone acetate in neoadjuvant therapy for surgically resectable high-risk or very high-risk prostate cancer after radical prostatectomy

SECONDARY OUTCOMES:
AEs/SAEs | Baseline up to 30 days after the last dose of study drug or before initiation of a new antitumor treatment, whichever occurred first
  The level of AEs defined by NCI-CTCAE v5.0. Safety assessments will be assessed and documented after initiation of study drug, regardless of relationship to study drug.
  The level of complications defined by Clavien-Dindo classification.
the 1-year PSA biochemical recurrence-free survival (bPFS) rate after radical prostatectomy in neoadjuvant therapy of paamiparib combined with abiraterone acetate in high- or very-high-risk prostate cancer | 3 years
  Defined as the proportion of patients who did not experience biochemical progression or death within 3 years of initiation of pamiparib treatment; biochemical progression was defined as an increase in serum PSA level to >0.2 ng/ml with 2 consecutive increases at least 3 months apart
Rate of Positive Surgical Margins | up to 8 months
  The proportion of subjects with positive surgical margins after radical prostatectomy
Downstaging rate of radical prostatectomy | four months to 2 years after surgery
  Downstaging rate of radical prostatectomy
Pathological response rate of neoadjuvant patients with HRR gene mutation | four months to 2 years after surgery
  Pathological response rate of neoadjuvant patients with HRR gene mutation
PSA response rate | up to 2 years
  The proportion of subjects with a ≥98% reduction in nadir PSA from baseline PSA during neoadjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: shun zhang, Dr., Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (2):
- China (2):
  - Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No